CLINICAL TRIAL: NCT00072449
Title: A Phase II Study Of Anti-CD20 Monoclonal Antibody (Rituximab) Therapy For Patients With Refractory Or Relapsed Primary CNS Lymphoma (PCNSL)
Brief Title: Rituximab in Treating Patients With Refractory or Relapsed Primary CNS Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual and lack of resources and priority due to combining 2 consortia
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NABTT-2201 CDR0000339737; U01CA062475 (NIH); NABTT-2201
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab

ARMS (1):
- Rituximab monotherapy (Experimental): Rituximab administered at a dose of 375mg/m2 as a single IV infusion every week for up to 8 weeks
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab in treating patients who have refractory or relapsed primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the radiographic response proportion in patients with refractory or recurrent primary CNS lymphoma treated with rituximab.

Secondary

* Determine the progression-free and overall survival of patients treated with this drug.
* Determine the toxicity profile of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV on days 1, 8, 15, and 22. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients may receive additional courses of rituximab off study at the discretion of the treating physician.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study within 5-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS lymphoma based on 1 of the following:

  * Histologically confirmed non-Hodgkin's B-cell lymphoma by brain biopsy or resection
  * Positive cerebrospinal fluid (CSF) cytology or immunohistochemical diagnosis of CSF monoclonality with or without measurable intracranial disease
  * Histologically confirmed vitreal lymphoma with measurable intracranial tumor
* CD20 positive by brain biopsy
* Measurable (greater than 1 cm in diameter) tumor by CT scan or MRI
* Progressed during first-line chemotherapy and/or radiotherapy OR relapsed after initial successful treatment
* No systemic lymphoma by CT scan of the chest, abdomen, and pelvis with contrast
* No leptomeningeal lymphoma by lumbar puncture for CNS cytology/flow cytometry
* No ocular lymphoma by slit lamp examination

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin less than 1.5 mg/dL
* Transaminases less than 4 times upper limit of normal

Renal

* Creatinine less than 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after study participation
* HIV negative
* Mini mental status examination score at least 15
* No concurrent serious infection
* No other medical illness that would preclude study treatment
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 90 days since prior biologic therapy
* No prior rituximab
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 3 months since prior radiotherapy

Surgery

* Not specified

Other

* Recovered from prior therapy
* More than 90 days since prior investigational drugs
* More than 90 days since prior use of a therapeutic device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-05; Primary Completion 2009-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, MD, MPH, Study Chair — Massachusetts General Hospital
Locations (9):
- United States (9):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Batchelor TT, Grossman SA, Mikkelsen T, Ye X, Desideri S, Lesser GJ. Rituximab monotherapy for patients with recurrent primary CNS lymphoma. Neurology. 2011 Mar 8;76(10):929-30. doi: 10.1212/WNL.0b013e31820f2d94. No abstract available. PMID 21383331

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab Monotherapy
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab Monotherapy
Number analyzed (Participants) | 12
Age Continuous [Median (Full Range); unit: years]
  age, years | 64 (31-81) [31 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Karnofsky Performance Status Scale [Median (Full Range); unit: Score] — 100 normal no complaints no disease 90 capable of normal activity few symptoms/disease 80 normal activity with some difficulty some symptoms or signs 70 caring for self not capable of normal activity or work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care and help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures or treatment 10 moribund rapidly progressive fatal disease processes 0 death
  Score | 85 [60 to 100]
Mini-Mental State Examination (MMSE) [Median (Full Range); unit: Score] — The mini-mental state examination (MMSE) is a 30-point questionnaire test used to screen for cognitive impairment. Commonly used to screen for dementia. It is also used to estimate the severity of cognitive impairment and to follow the course of cognitive changes in an individual over time. The MMSE test includes simple questions and problems in a number of areas: the time and place of the test, repeating lists of words, arithmetic such as the serial sevens, language use and comprehension, and basic motor skills. The Higher your score, the higher your function.
  Score | 29 [18 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response
Description: it at any time point patient progresses no more scans are required, patient is off study
Time Frame: 1 month, 2 months and then q3months
Measure: Number; unit: participants
Arm/Group | Rituximab Monotherapy
Number analyzed (Participants) | 11
participants | 4

2. Secondary Outcome: Progression-free Survival
Description: pt had MRI every 3 months
Time Frame: pt had MRI q3months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab Monotherapy
Number analyzed (Participants) | 12
days | 57 [29 to 175]

3. Secondary Outcome: Overall Survival
Description: survival was evaluated q 2months
Time Frame: 47 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab Monotherapy
Number analyzed (Participants) | 12
months | 20.9 [2.9 to 47]

4. Secondary Outcome: Toxicity
Description: patients only received drug for 8 weeks
Time Frame: 8 weeks - 2 cycles
Measure: Number; unit: related episodes
Arm/Group | Rituximab Monotherapy
Number analyzed (Participants) | 12
related episodes | 4

ADVERSE EVENTS:
Time Frame: While on active treatment and for on month after treatment, which meant 8 weeks of active treatment and 1 month follow-up.
Description: Note that not all AEs are related to treatment
Arm/Group | Rituximab Monotherapy
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Monotherapy (N=12)
infection-sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Monotherapy (N=12)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
"Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip)" (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Ataxia (incoordination) (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 2 (2)
"Constitutional Symptoms - Other (Specify, cold (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema: limb (General disorders) | 4 (6)
"Fatigue (asthenia, lethargy, malaise)" (General disorders) | 9 (9)
"Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)" (General disorders) | 1 (1)
Gastrointestinal-other - mouth sores (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
"Infection - Other (Specify, __)" - oral thrush (Infections and infestations) | 1 (1)
"Infection - Other (Specify, __)" - shingles (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mood alteration - Anxiety (Psychiatric disorders) | 3 (3)
Mood alteration - Depression (Psychiatric disorders) | 1 (1)
"Muscle weakness, generalized or specific area (not due to neuropathy) - Left-sided" (Musculoskeletal and connective tissue disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 2 (2)
Neuropathy: cranial - CN II Vision (Eye disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 2 (3)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pain - Back (Injury, poisoning and procedural complications) | 1 (1)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Head/headache (Nervous system disorders) | 4 (4)
Pain - Miuscle (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
"Phosphate, serum-low (hypophosphatemia)" (Metabolism and nutrition disorders) | 1 (1)
Platelets (Investigations) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
"Pulmonary/Upper Respiratory - Other (Specify, __)" (Respiratory, thoracic and mediastinal disorders) | 1 (1) — diminished breath sounds
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rigors/chills (General disorders) | 3 (3)
seizure (Nervous system disorders) | 1 (1)
somnolence (Nervous system disorders) | 1 (1)
speech impairment (Nervous system disorders) | 2 (2)
thrombosis (Vascular disorders) | 1 (1) — RLE DVT
tinnitus (Ear and labyrinth disorders) | 1 (1)
tremor (Nervous system disorders) | 1 (1)
vision blurred (Eye disorders) | 3 (3)
vomiting (Gastrointestinal disorders) | 2 (2)
Alkaline phosphatase (Investigations) | 2 (2)
Creatinine (Investigations) | 1 (1)
hemoglobin (Investigations) | 6 (21)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (9)
platelets (Infections and infestations) | 4 (8)
aspartate aminotransferase SGOT (Infections and infestations) | 3 (3)
alanine aminotransferase SGPT (Investigations) | 3 (5)
total bilirubin (Investigations) | 1 (1)
white blood count (Blood and lymphatic system disorders) | 2 (8)

LIMITATIONS AND CAVEATS:
Study terminated early due to slow accrual and lack of resources and priority due to NCI mandate of combining two consortia. Unable to fully analyze the data, or objectives, not enough patients. Not able to do statistics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No